CLINICAL TRIAL: NCT00902265
Title: Efficacy and Safety of Nocturin 0.1 mg Tablets in Treatment of Nocturia in Patients With Nocturnal Polyuria, Lower Urinary Tract Symptoms (LUTS) and Benign Prostate Syndrome (BPS).
Brief Title: Efficacy and Safety of Desmopressin (Nocturin®) 0.1 mg Tablets in Treatment of Nocturia in Participants With Benign Prostate Syndrome (BPS)
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Other Study IDs: FE992026 CS33
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Results first posted 2011-04-11 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Nocturia Associated With Nocturnal Polyuria
MeSH Terms: interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- desmopressin: Participants with benign prostate syndrome suffering from nocturia associated with nocturnal polyuria.
  Drug given by prescription.
  Interventions: Drug: desmopressin

INTERVENTIONS:
Drug: desmopressin — desmopressin (Nocturin®) 0.1 mg tablet per day for 12 weeks
  Other Names: Nocturin®

SUMMARY:
Documentation of the efficacy and safety of desmopressin (Nocturin®) 0.1 mg tablet. Observation of patients with benign prostate syndrome, in whom nocturia associated with nocturnal polyuria is treated with desmopressin (Nocturin®) 0.1 mg tablet focusing on number of nocturnal voids, ratio of night/24-h urine volume (%), duration of first undisturbed sleep period and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Therapeutic need according to Summary of Product Characteristics
* Written informed consent

Exclusion Criteria:

* Contraindications according to Summary of Product Characteristics

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: private practices
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2009-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (140):
- Germany (140):
  - Investigational Site - Pauwelsstraße 30, Aachen
  - Investigational Site - Sanatoriumstraße 10, Aachen
  - Investigational Site, Arnsberg
  - Investigational Site, Bad Bergzaben
  - Investigational Site, Bad Schönborn
  - Investigational Site, Baierbrunn
  - Investigational Site, Bergisch Gladbach
  - Investigational Site - Breite Straße 37, Berlin
  - Investigational Site - Britzer Damm 63, Berlin
  - Investigational Site - Florastraße 44, Berlin
  - Investigational Site - Fritz-Reuter-Straße 6-8, Berlin
  - Investigational Site - Heerstraße 435, Berlin
  - Investigational Site - Kaiserdamm 12, Berlin
  - Investigational Site - Kurfürstendamm 33, Berlin
  - Investigational Site - Marburger Straße 12/13, Berlin
  - Investigational Site - Mehrower Allee 22, Berlin
  - Investigational Site - Rüdesheimer Straße 43, Berlin
  - Investigational Site - Schnellerstraße 123, Berlin
  - Investigational Site - Tempelhofer Damm 214, Berlin
  - Investigational Site - Turmstraße 82, Berlin
  - Investigational Site, Biberach
  - Investigational Site, Bochum
  - Investigational Site, Bonn
  - Investigational Site - Friedrich-Wilhelm-Str. 43/44, Braunschweig
  - Investigational Site - Güldenstraße 19-20, Braunschweig
  - Investigational Site - Humboldtstraße 4, Braunschweig
  - Investigational Site - Küchenstraße 10, Braunschweig
  - Investigational Site - Ritterbrunnen 7, Braunschweig
  - Investigational Site - Dr.-Franz-Mertens-Str. 8, Bremerhaven
  - Investigational Site - Georgstraße 44, Bremerhaven
  - Investigational Site, Bruchköbel
  - Investigational Site, Brühl
  - Investigational Site, Butzbach
  - Investigational Site, Bückeburg
  - Investigational Site, Büdingen
  - Investigational Site - Großer Plan 11, Celle
  - Investigational Site - Neumarkt 1d, Celle
  - Investigational Site - Hohenstaufenring 59, Cologne
  - Investigational Site - Wilhelm-Ewald-Weg 1, Cologne
  - Investigational Site - Zeppelinstraße 1, Cologne
  - Investigational Site, Cottbus
  - Investigational Site, Dorsten
  - Investigational Site - Hansastraße 14-16, Dortmund
  - Investigational Site - Markt 4, Dortmund
  - Investigational Site - Wittbräucker Str. 2, Dortmund
  - Investigational Site, Düsseldorf
  - Investigational Site, Eilenburg
  - Investigational Site, Eisenberg
  - Investigational Site, Eisleben Lutherstadt
  - Investigational Site, Erftstadt
  - Investigational Site - Altessener Str. 400a, Essen
  - Investigational Site - Gerichtsstraße 32, Essen
  - Investigational Site - Humannstraße 3, Essen
  - Investigational Site - Rüttenscheider Stern 5, Essen
  - Investigational Site - Bologarostraße 131, Frankfurt a.M.
  - Investigational Site - Eschersheimer Landstr. 544, Frankfurt a.M.
  - Investigational Site - Oeder Weg 72, Frankfurt a.M.
  - Investigational Site - Ginnheimer Landstraße 88, Frankfurt am Main
  - Investigational Site, Gardelegen
  - Investigational Site - Zum Ehrenmal 21, Gelsenkirchen
  - Investigational Site, Gera
  - Investigational Site, Gifhorn
  - Investigational Site, Gotha
  - Investigational Site, Grimma
  - Investigational Site - Diesterwegstraße 39, Halle
  - Investigational Site - Nimeyerstraße 23, Halle
  - Investigational Site - Grindelberg 3, Hamburg
  - Investigational Site - Möllner Landstraße 27, Hamburg
  - Investigational Site, Hanover
  - Investigational Site, Hemmoor
  - Investigational Site, Homburg
  - Investigational Site, Höchheim
  - Investigational Site, Hönow
  - Investigational Site - Dornburger Straße 17a, Jena
  - Investigational Site - Ernst-Abbe-Platz 3-4, Jena
  - Investigational Site - Zitzmannstraße 2, Jena
  - Investigational Site, Kaiserslautern
  - Investigational Site, Kamp-Lintfort
  - Investigational Site, Karlsruhe
  - Investigational Site, Kiel
  - Investigational Site, Kleinmanchow
  - Investigational Site, Köln-Zollstock
  - Investigational Site, Königs Wusterhausen
  - Investigational Site, Königswinter
  - Investigational Site, Lahr
  - Investigational Site, Landau/Isar
  - Investigational Site, Landshut
  - Investigational Site, Langenau
  - Investigational Site, Lauterbach
  - Investigational Site, Leipzig
  - Investigational Site, Lindau
  - Investigational Site, Magdeburg
  - Investigational Site, Marburg
  - Investigational Site, Markkleeberg
  - Investigational Site, Meschede
  - Investigational Site, Nettetal
  - Investigational Site, Neunkirchen
  - Investigational Site, Nienburg
  - Investigational Site, Norderstedt
  - Investigational Site - August-Bebel-Platz 33-34, Nordhausen
  - Investigational Site - Bahnhofstraße 17, Nordhausen
  - Investigational Site - Bahnhofstraße 8, Nordhausen
  - Investigational Site, Offenbach
  - Investigational Site, Offenburg
  - Investigational Site, Oldenburg
  - Investigational Site, Porta Westfalica
  - Investigational Site - Allee nach Sanssouci 7, Potsdam
  - Investigational Site - Großbeerenstraße 301, Potsdam
  - Investigational Site, Quakenbrück
  - Investigational Site, Quedlinburg
  - Investigational Site, Recklinghausen
  - Investigational Site - Materialhofstraße 9-11, Rendsburg
  - Investigational Site, Ribnitz-Damgarten
  - Investigational Site, Rinteln
  - Investigational Site, Rostock
  - Investigational Site - Berliner Promenade 15, Saarbrücken
  - Investigational Site - Kaiserslauterer Str. 26, Saarbrücken
  - Investigational Site - Heckenstraße 10, Salzgitter
  - Investigational Site - In den Blumentriften 62, Salzgitter
  - Investigational Site, Salzmünde
  - Investigational Site, Schleswig
  - Investigational Site - Am Ostentor 5, Schwerte
  - Investigational Site - Karl-Gerharts-Straße 2, Schwerte
  - Investigational Site, Seehausen
  - Investigational Site, Solingen
  - Investigational Site, Sömmerda
  - Investigational Site, Taucha
  - Investigational Site, Teltow
  - Investigational Site, Tostedt
  - Investigational Site - Fleischstraße 20, Trier
  - Investigational Site - Kutzbachstraße 7, Trier
  - Investigational Site - Einsteinstraße 59, Ulm
  - Investigational Site - Olgastraße 103, Ulm
  - Investigational Site - Olgastraße 139, Ulm
  - Investigational Site, Velbert
  - Investigational Site, Wesel
  - Investigational Site, Wilhelmshaven
  - Investigational Site, Witten
  - Investigational Site - Langerfelder Straße 115, Wuppertal
  - Investigational Site - Morianstraße 10, Wuppertal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a post marketing, non-randomized surveillance study. The 138 participants were screened from 60 German sites.
  The study planned for two visits - baseline (week 0 and week 12). Participants could opt for an optional visit between week 0 and week 12 (17 participants did not opt for optional visit).
Groups:
- Desmopressin 0.1 mg: Participants with benign prostate syndrome suffering from nocturia associated with nocturnal polyuria.
  Drug given by prescription.
Period: Overall Study
Arm/Group | Desmopressin 0.1 mg
Started | 138
Participants Who Received Treatment | 137
Completed | 132
Not Completed | 6
Not completed — Lost to Follow-up Prior to First Visit | 1
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Desmopressin 0.1 mg
Number analyzed (Participants) | 137
Age Continuous [Mean (Standard Deviation); unit: years] | 62.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 137
Region of Enrollment [Number; unit: participants]
  Germany | 137

OUTCOME MEASURES:

1. Primary Outcome: Overall Mean Change From Baseline in Mean Number of Nighttime Voids at Week 12
Description: The number of nighttime voids was calculated over 48-hours period prior to baseline and week 12 visits. Calculated as Week 12 measure - Baseline measure.
Time Frame: Baseline, Week 12
Population: Intent to treat (ITT) population --All participants who received at least one dose of study drug and provided at least one primary efficacy measure (i.e., number of nocturnal voids)
Measure: Mean (Standard Deviation); unit: Number of nocturnal voids
Arm/Group | Desmopressin 0.1 mg
Number analyzed (Participants) | 132
Number of nocturnal voids | -2.01 (1.13)

2. Secondary Outcome: Mean Change From Baseline in Ratio of Nighttime Urine Volume to 24-hour Urine Volume at Week 12
Description: The ratio of nighttime urine volume to 24-hour urine volume is calculated as the urine volume (volume of all voids after going to bed plus the first morning void) / 24-hour urine volume. Ratios are calculated at baseline and week 12 and difference between the two time points is reported here.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Desmopressin 0.1 mg
Number analyzed (Participants) | 114
ratio | -14.0 (11.9)

3. Secondary Outcome: Mean Change From Baseline in Initial Period of Undisturbed Sleep at Week 12
Description: Initial period of undisturbed sleep is calculated as the number of hours between falling asleep and waking for the first time during the night to void. Change is calculated at Week 12 - baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Desmopressin 0.1 mg
Number analyzed (Participants) | 124
Hours | 1.69 (1.16)

4. Secondary Outcome: Mean Change From Baseline of Total International Prostate Symptom Score (IPSS) at Week 12
Description: The International Prostate Symptoms Score (IPSS) is a self-administered 8 item questionnaire designed to assess urination frequency and Quality of Life (QOL). The first 7 items are summed into a total score and question urination frequency. They are scaled 0-5, with higher numbers indicating greater severity of symptoms. The last question (item 8) concerns QOL and is scaled 0-6 where higher numbers indicate lower quality of life due to symptoms. The total scale across all questions is 0-41, with higher scores representing worse symptoms.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Desmopressin 0.1 mg
Number analyzed (Participants) | 131
Units on a scale | -4.86 (4.22)

5. Secondary Outcome: Mean Change From Baseline International Prostate Symptom Score (IPSS) Quality of Life Score at Week 12
Description: The International Prostate Symptoms Score (IPSS) is a self-administered 8 item questionnaire designed to assess urination frequency and Quality of Life (QOL). The last question (item 8) concerns Quality of Life (QOL) and is scaled 0-6 where higher numbers indicate lower quality of life due to symptoms. Higher scores represent worse Quality of Life (QoL).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Desmopressin 0.1 mg
Number analyzed (Participants) | 117
Units on a scale | -1.56 (1.05)

6. Secondary Outcome: Mean Change From Baseline in Total Score in Leeds Sleep Evaluation Questionnaire (LSEQ) at Week 12
Description: The LSEQ is a self-administered 10-item visual analog scale questionnaire designed to assess sleep quality. The 10 individual items are scored 1 to 100, with the total score ranging from 0 - 1,000. Higher numbers indicate lower sleep quality.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Desmopressin 0.1 mg
Number analyzed (Participants) | 129
Units on a scale | -15.1 (12.1)

7. Secondary Outcome: Change From Baseline in Degree of Bother Due to Frequency of Daytime Voiding Assessed by The International Consultation on Incontinence Modular Questionnaire - Nocturia (ICIQ-N)
Description: The ICIQ-N is a self-administered 4-item questionnaire designed to assess the frequency and bother of daytime and nighttime urination. In questions 1 and 2 participants were asked to estimate the frequency of both daytime voiding (all voids before going to bed excluding the first morning void) and rate the degree of bother of daytime urination on a scale ranging from 0 (not at all) to 10 (a great deal). Higher numbers indicate lower Quality of Life (QoL).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Desmopressin 0.1 mg
Number analyzed (Participants) | 127
Units on a scale | -2.25 (2.25)

8. Secondary Outcome: Change From Baseline in Degree of Bother Due to Frequency of Nighttime Voiding Assessed by The International Consultation on Incontinence Modular Questionnaire - Nocturia (ICIQ-N)at Week 12
Description: The ICIQ-N is a self-administered 4-item questionnaire designed to assess the frequency and bother of daytime and nighttime urination. In questions 3 and 4, participants were asked to estimate the frequency of nighttime voiding (number of voids after going to bed plus the first morning void) and rate the degree of bother of nighttime urination on a scale ranging from 0 (not at all) to 10 (a great deal). Higher numbers indicate lower Quality of Life (QOL).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Desmopressin 0.1 mg
Number analyzed (Participants) | 129
Units on a scale | -4.00 (2.49)

9. Secondary Outcome: Participants With Treatment Emergent Adverse Events (AEs)
Time Frame: Week 1 to Week 12
Population: Safety Population, consisting of participants who took at least one dose of desmopressin
Measure: Number; unit: Participants
Arm/Group | Desmopressin 0.1 mg
Number analyzed (Participants) | 137
Participants
  All Adverse Events | 3
  Deaths | 0
  Serious Adverse Events | 0
  AEs Leading to Discontinuation | 2

ADVERSE EVENTS:
Arm/Group | Desmopressin 0.1 mg
Serious Adverse Events (participants affected / at risk) | 0/137
Other Adverse Events (participants affected / at risk) | 0/137

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI gives Ferring a draft manuscript 30 days before submission for the final form for to any journal for review and comments. Ferring can ask that confidential information be removed.